CLINICAL TRIAL: NCT03170427
Title: Impedance Cardiography as Tool for Continuous Hemodynamic Monitoring During Cesarean Section: Randomized, Prospective Double Blind Study
Brief Title: Impedance Cardiography as Tool for Continuous Hemodynamic Monitoring During Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Foggia (Other)
Responsible Party: Principal Investigator, Cotoia Antonella, researcher, University of Foggia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 18/CE/2012
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Cardiography, Impedance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 mg (2 mL) levobupivacaine (Sham Comparator): 8mg (2ml) levobupivacaine plus 20 µg fentanyl will be given intrathecally by spinal anesthesia. The impendance cardiography, the sensory and motor block will be monitored
  Interventions: Device: Impedance cardiography; Diagnostic Test: Sensory levels; Diagnostic Test: Motor block; Diagnostic Test: Sensory level
- 6 mg (1.6 mL) levobupivacaine (Active Comparator): 6mg (1.6ml) levobupivacaine plus 20 µg fentanyl will be given intrathecally by spinal anesthesia. The impendance cardiography, the sensory and motor block will be monitored
  Interventions: Device: Impedance cardiography; Diagnostic Test: Sensory levels; Diagnostic Test: Motor block; Diagnostic Test: Sensory level

INTERVENTIONS:
Device: Impedance cardiography — hemodynamic variation measured by impedance cardiography in healthy pregnant undergoing to cesarean section treated with 8mg or 6mg of levobupivacaine
Diagnostic Test: Sensory levels — Sensory levels are checked using ice test cold
Diagnostic Test: Motor block — motor block is measured by modified Bromage scale
Diagnostic Test: Sensory level — Sensory levels are checked using touch with alcohol puffs

SUMMARY:
Impedance Cardiography (ICG) is a non-invasive tool for continuous hemodynamic monitoring. Aims of our study is to assess the utility of ICG to evaluate the hemodynamic impact of 6 mg (GL6) vs 8 mg (GL8) levobupivacaine combined with fentanyl in healthy patients undergoing elective cesarean section; secondary, to compare the duration and quality of analgesia and anesthesia

DETAILED DESCRIPTION:
On arrival in the recovery room the ICG non-invasive blood pressure cuff will be placed on the left arm, two sensors will be placed above the clavicle on each side of the neck, and two sensors will bw placed on either side of the thorax at midaxillary line corresponding to the level of the xiphoid process. Using a computer- generated sequence of numbers, patients will be randomly allocated in one of the two groups: 6 mg (1.6 mL) levobupivacaine + 20 µg fentanyl (GL6 group) or 8 mg (2 mL) levobupivacaine + 20 µg fentanyl (GL8 group). Continuous spinal epidural anesthesia (CSE) will be performed with patient in sitting position: a 18-gauge Tuohy needle will be inserted into the L2-L3 interspace using the loss of resistance of saline technique to identify the epidural space; a 27-gauge Withacre spinal needle will be then placed through the Tuohy needle until the dura mater wwill be punctured and isobaric undiluted levobupivacaine plus 20 µg fentanyl was administered. Afterwards, an epidural catheter (Espocan, B.Braun, Melsungen, Germany) wwill be inserted 4 cm into the epidural space.

ELIGIBILITY:
Inclusion Criteria:

* pregnant undergoing elective Caesarean delivery at term of singleton pregnancy, with American Society of Anesthesiologists physical status of class I or II, without preeclampsia or diabetes,

Exclusion Criteria:

* Patient with a known allergy to amide local anesthetics and other drugs, with BMI≥40 kg/m2, cardiologic or systemic disease, in treatment with antihypertensive or anticoagulant

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2014-05-31 (Actual)

PRIMARY OUTCOMES:
hemodynamic continuous monitoring by impedance cardiography | intraoperative time
  Impedance cardiography as a tool for hemodynamic monitoring during cesarean section

SECONDARY OUTCOMES:
onset of sensory block | intraoperative time
  onset time of sensory block after intrathecal levobupivacaine
offset of sensory block | intraoperative time
  offset time of sensory block after intrathecal levobupivacaine
onset of motor block | intraoperative time
  onset time of motor block after intrathecal levobupivacaine
offset of motor block | intraoperative time
  offset time of motor block after intrathecal levobupivacaine

REFERENCES:
- [Derived] D'Ambrosio A, Cotoia A, Beck R, Salatto P, Zibar L, Cinnella G. Impedance cardiography as tool for continuous hemodynamic monitoring during cesarean section: randomized, prospective double blind study. BMC Anesthesiol. 2018 Mar 27;18(1):32. doi: 10.1186/s12871-018-0498-4. PMID 29587655